CLINICAL TRIAL: NCT02913235
Title: Does Short Term Discontinuation of Self-performed Oral Hygiene Procedures Influence the Composition of the Salivary Microbiota?
Brief Title: Salivary Bacterial Associations to Short Term Discontinuation of Self-performed Oral Hygiene
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: The Forsyth Institute (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Daniel Belstrøm, DDS, PhD, Assistant professor, University of Copenhagen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UCPH_OI_002
Record Dates: First submitted 2016-09-20; First posted 2016-09-23 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Mouth Diseases
Keywords: biofilm; saliva; bacteria; oral hygiene
MeSH Terms: conditions — Mouth Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oral hygiene discontinuation group (Experimental): The intervention of the present study is discontinuation of regular oral hygiene procedures for a period of 10 days. Discontinuation of oral hygiene will allow undisturbed biofilm formation (supragingival dental plaque) along the gingival margin of the teeth. After 10 days all individuals will resume regular oral hygiene. Clinical registrations and collection of microbiological samples (supragingival and saliva) will be performed at baseline and 4, 7 and 10 days after discontinuation of regular oral hygiene, and will be repeated 14 days after regular oral hygiene has been resumed.
  Interventions: Procedure: Oral hygiene discontinuation group

INTERVENTIONS:
Procedure: Oral hygiene discontinuation group — Discontinuation of regular oral hygiene for 10 days

SUMMARY:
The purpose of the present investigation is to record and compare bacterial compositions in supragingival plaque samples and saliva samples in subjects discontinuing regular oral hygiene for 10 days. The hypothesis is that the composition of the salivary microbiota might reflect local bacterial alterations in relation to discontinuation of oral hygiene.

DETAILED DESCRIPTION:
35 orally healthy individuals will be enrolled in this study, in which they will discontinue regular oral hygiene procedures for a period of 10 days. Clinical registrations and collection of microbiological samples (supragingival and saliva) will be performed at baseline and 4, 7 and 10 days after discontinuation of regular oral hygiene, and will be repeated 14 days after regular oral hygiene has been resumed.

ELIGIBILITY:
Inclusion Criteria:

* Oral and systemically healthy individuals

Exclusion Criteria:

* Periodontitis
* Dental caries
* Systemic diseases or medications with known associations to oral health
* Antibiotics within the latest 6 month

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-09; Primary Completion 2017-01-02 (Actual); Study Completion 2017-01-02 (Actual)

PRIMARY OUTCOMES:
Comparison of changes in α-diversity in saliva samples before and after discontinuation of regular oral care | 10 days of discontinuation of regular oral care and 14 days after resuming regular oral care
  Comparison of α-diversity in saliva samples before and after discontinuation of regular oral hygiene

SECONDARY OUTCOMES:
Comparison of species specific changes in saliva samples before and after discontinuation of regular oral care | 10 days of discontinuation of regular oral care and 14 days after resuming regular oral care
  Comparison of relative abundance of bacterial species in saliva samples at baseline to samples collected 10 days after discontinuation of regular oral hygiene and to samples collected 14 days after oral hygiene procedures has been resumed

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Belstrøm, DDS, PhD, Principal Investigator — University of Copenhagen

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Belstrom D, Sembler-Moller ML, Grande MA, Kirkby N, Cotton SL, Paster BJ, Twetman S, Holmstrup P. Impact of Oral Hygiene Discontinuation on Supragingival and Salivary Microbiomes. JDR Clin Trans Res. 2018 Jan;3(1):57-64. doi: 10.1177/2380084417723625. Epub 2017 Jul 31. PMID 29662960